CLINICAL TRIAL: NCT00575029
Title: Evaluation of the Time Course of Adrenal Suppression and Adrenal Recovery After Ingestion of Megestrol Acetate
Brief Title: Adrenal Suppression and Adrenal Recovery Induced by Megestrol Acetate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Donald Bodenner MD, university of arkansas for medical sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 26835
Record Dates: First submitted 2007-12-13; First posted 2007-12-17 (Estimated); Results first posted 2011-08-29 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2011-07

CONDITIONS: Adrenal Insufficiency
Keywords: megestrol acetate; adrenal insufficiency; adrenal suppression
MeSH Terms: conditions — Adrenal Insufficiency | interventions — Megestrol Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- megace treatment (Experimental): Study subjects will be given 600mg of MA for oral ingestion per day for duration of 8 weeks. They will be monitored every week clinically for the development of adrenal insufficiency by review of symptoms, physical exam, body weight, pulse, and blood pressure. Subjects also will undergo biochemical evaluation of adrenal status every two weeks by measurement of serum electrolytes, serum cortisol, serum adrenocorticotropic hormone(ACTH) levels, and the adrenal response to a low dose ACTH (1µgm) stimulation test(see methods).
  Interventions: Drug: megestrol acetate

INTERVENTIONS:
Drug: megestrol acetate — 600 mg by mouth daily

SUMMARY:
Megestrol Acetate (MA) is a progesterone-like hormone that has been utilized as a birth control agent, chemotherapeutic drug, and more recently, to induce appetite and weight gain in patients malnourished as a result of radiation therapy, chemotherapy, cystic fibrosis, AIDS, or dementia. The mechanism of MA-stimulated appetite and weight gain is unknown.

Although only approved to combat weight loss associated with AIDS and cancer, MA is frequently prescribed for long periods of time to prevent or reverse weight loss in nursing home residents and in elderly patients with serious illnesses in the community. Little data is available to support this practice. Among its many properties, MA acts as a partial glucocorticoid agonist, and long term and short term use of MA may results in adrenal suppression. The rapidity of the onset of MA-induced adrenal suppression and the time course of resumption of normal adrenal function after discontinuation of MA is completely unknown. As a consequence, it is unclear whether MA can be given safely for short periods of time or whether glucocorticoid administration is necessary after abruptly stopping MA treatment. The increased use of MA in the frail elderly, where even partial adrenal insufficiency may pose a substantial risk of adrenal crisis after an illness, requires a clear understanding of these issues. To address these concerns, we will evaluate adrenal function before, during, and after MA administration in healthy volunteers between the ages of 60 and 85 years.

ELIGIBILITY:
Inclusion Criteria:

* Elderly males and females
* Age 65-80 years
* With stable (no history of urgent/ emergent care visits with health care provider/s in the preceding 2 months), medical conditions

Exclusion Criteria:

Subjects will be excluded if they have a history of (H/O):

* Dementia
* Adrenal disease
* Thromboembolism
* Diabetes mellitus
* Liver disease
* Electrolyte abnormalities; or
* Vaginal bleeding
* Hypertriglyceridemia
* CAD with CHF
* Unstable depression
* Schizophrenia; and
* Morbidly obese subjects.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 7 (Actual)
Dates: Start 2004-04; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: donald l bodenner, Principal Investigator — associate professor
Locations (1):
- University of Arkansas For Medical Sciences, Little Rock, Arkansas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment 4/04 to 7/04.
Groups:
- Megestrol Acetate: Study subjects will be given 600mg of MA (megestrol acetate) for oral ingestion per day for duration of 8 weeks.
Period: Overall Study
Arm/Group | Megestrol Acetate
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Megestrol Acetate
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 7
Age Continuous [Mean (Standard Deviation); unit: years] | 68 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adrenal Insufficiency
Description: Number of participants with adrenal insufficiency after treatment with megestrol acetate assessed by ACTH stimulated cortisol levels less than normal (21 ug/dl) measured weekly for 8 weeks or when adrenal insufficiency is clinically encountered
Time Frame: stimulated acth stimulated cortisol levels weekly for 8 weeks or until adrenal insufficiency is encountered
Measure: Number; unit: participants
Arm/Group | Megestrol Acetate
Number analyzed (Participants) | 7
participants | 7

2. Primary Outcome: Time Required for Recovery From Adrenal Suppression to Normal Adrenal Function
Description: the number of weeks required for participants to recover from adrenal suppression as assessed by a normal ACTH stimulation test (cortisol level >21 mcg/dl)
Time Frame: weekly for up to 6 weeks
Measure: Number; unit: weeks
Arm/Group | Megestrol Acetate
Number analyzed (Participants) | 7
weeks
  participant 1 | 6
  participant 2 | 2
  participant 3 | 2
  participant 4 | 2
  participant 5 | 2
  participant 6 | 2
  participant 7 | 2

ADVERSE EVENTS:
Arm/Group | Megestrol Acetate
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

LIMITATIONS AND CAVEATS:
funding became an issue limiting the number of patients enrolled

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes